CLINICAL TRIAL: NCT00304707
Title: Bupropion Treatment for Smokers in Recovery
Brief Title: Effectiveness of Bupropion for Smokers Recovering From Alcohol Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, David Kalman, Principal Investigatgor, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA017370 (NIH); R01DA017370 (NIH)
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Smoking Cessation; Alcohol-Related Disorders
MeSH Terms: conditions — Smoking Cessation; Alcohol-Related Disorders | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 2 (Experimental): participants in this arm receive bupropion
  Interventions: Drug: Bupropion
- 1 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bupropion — 300 mg QD
  Arms: 2
Drug: placebo — placebo
  Arms: 1

SUMMARY:
Smoking is often a problem for alcohol dependent individuals. Many people who seek treatment for alcohol dependence are unable to quit smoking. The purpose of this study is to evaluate the effectiveness of bupropion, an antidepressant medication, in treating smokers receiving treatment for alcohol dependence.

DETAILED DESCRIPTION:
Past research suggests that over 75% of alcohol dependent individuals in early alcohol recovery smoke cigarettes; smoking-related mortality exceeds alcohol-related mortality in this population. Many alcohol dependent individuals in early recovery are interested in smoking cessation treatment; however, studies indicate that these smokers find it very difficult to quit smoking. More effective treatment methods are needed for smokers in early alcohol recovery. Bupropion is a dopaminergic antidepressant that may be effective in treating nicotine dependent individuals. The purpose of this study is to evaluate the effectiveness of bupropion in nicotine dependent individuals receiving treatment for alcohol dependence. In addition, this study will investigate the psychological mechanisms that may mediate the efficacy of bupropion in smoking cessation. We will also collect DNA from subjects in order to explore whether response to bupropion is mediated by particular genetic variants in the dopaminergic, metabolic and nicotinic receptor systems of smokers.

Participants will be randomly assigned to receive either 300 mg of bupropion or placebo, daily for 8 weeks. In addition, all participants will receive a nicotine patch for 7 weeks. This will consist of a 21-mg nicotine patch for 4 weeks, a 14-mg nicotine patch for 2 weeks, and a 7-mg nicotine patch for 1 week. All participants will undergo seven counseling sessions. Follow-up visits will occur at Weeks 7, 12, and 24. Pre-quit variables (e.g., smoking satisfaction) and three post-quit variables (craving, nicotine withdrawal, and negative effects) will be evaluated at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* Smokes a minimum of 10 cigarettes daily for at least 1 year prior to study entry
* Abstinence from alcohol and other non-nicotine drugs for between 1 and 12 months at time of study entry
* Meets criteria for alcohol dependence or abuse in the 12 months prior to study entry

Exclusion Criteria:

* History of seizures, head trauma and/or severe hepatic cirrhosis
* Current use of medications known to affect smoking behavior and/or cessation
* Use of tricyclic antidepressant medication and monoamine oxidase inhibitors
* Major depressive disorder within the month prior to study entry
* Eating disorder within the year prior to study entry
* History of bipolar or psychotic disorder
* Pregnant or breastfeeding
* Unstable serious medical disorder
* History of migraines
* Currently using smokeless tobacco, pipes, or cigars

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2005-04; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kalman, PhD, Principal Investigator — Boston University
Locations (1):
- ENRM Veterans Hospital, Bedford, Massachusetts, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion 300-mg Capsules: participants in this arm receive bupropion
  Bupropion: 300 mg QD
Period: Overall Study
Arm/Group | Bupropion 300-mg Capsules | Placebo
Started | 73 | 70
Completed | 66 | 64
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion 300-mg Capsules | Placebo | Total
Number analyzed (Participants) | 73 | 70 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (7.5) | 47.8 (10.5) | 48.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 58 | 59 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 16 | 36
  White | 53 | 54 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 73 | 70 | 143

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence
Description: The number of subjects in each treatment group who were smoking abstinent (7-day point prevalence) at week 7 (end of treatment), week 11 and week 24.
Time Frame: week 7, week 11 and week 24 after scheduled quit day
Measure: Number; unit: participants
Arm/Group | Bupropion 300-mg Capsules | Placebo
Number analyzed (Participants) | 73 | 70
participants
  week 7 | 19 | 21
  week 11 | 12 | 9
  week 24 | 6 | 11

ADVERSE EVENTS:
Arm/Group | Bupropion 300-mg Capsules | Placebo
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/70
Other Adverse Events (participants affected / at risk) | 7/73 | 2/70
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bupropion 300-mg Capsules (N=73) | Placebo (N=70)
insomnia (Nervous system disorders) | 5 | 2
Dry mouth (Endocrine disorders) | 2 | 1
Rise in systolic blood pressure (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No